CLINICAL TRIAL: NCT00073606
Title: Intraspinal Plasticity Associated With Locomotor Learning
Brief Title: Spinal Cord Plasticity
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040054; 04-N-0054
Record Dates: First submitted 2003-12-01; First posted 2003-12-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-05-20

CONDITIONS: Healthy
Keywords: Spinal Reflexes; Locomotion; Motor Practice; Healthy Volunteer; HV

SUMMARY:
This study will examine the role of the spinal cord in improving leg movements after physical training in healthy people. The results of this study may be helpful in developing new rehabilitation therapies for people with impaired leg function.

Healthy volunteers between 21 and 65 years of age may be eligible for this study. Candidates will be screened with a brief medical history and physical examination.

Participants will undergo EMG-H reflex measurement while pedaling on a stationary bicycle. For this test, the subject is given an electrical stimulation at the nerve at the back of the knee while pedaling on a stationary bicycle. The shock produces a jerky movement called the "H reflex." The muscular activity causing these reflexes is measured using electrodes (small metal disks) filled with a conductive gel and taped to the skin over the calf muscle. The nerve is stimulated at four different frequencies during the experiment. While cycling, pedal resistance changes, making it harder or easier to pedal.

On study day 1, participants have EMG-H reflex measurement to determine baseline performance, then a training session to prepare for the actual test, and then a post-training test to measure performance again. The test is repeated on days 2, then between days 5 and 8, and again between days 11 and 14. The screening and first visit last 2 hours; the remaining test visits are 1 hour each. The bicycling time is only 15 minutes during training and 5 minutes at each test session.

DETAILED DESCRIPTION:
Objectives

We aim to determine whether the development of a motor memory in the human spinal cord circuitry (expressed as a down regulation of the monosynaptic soleus H reflex) after a brief period of learning of a locomotor skill, is intrinsically encoded at the spinal cord level or if it is determined by descending suprasegmental influences.

The results of this study would be useful for designing new rehabilitation strategies based upon manipulation of peripheral inputs aimed at activating spinal cord circuitry for motor recovery independent of the higher centers.

Study population

Seventy (70) healthy volunteers (median age 21-65) will participate in the study.

Design

Subjects will complete one training session (using a recumbent cycle ergometer) and will be tested physiologically and behaviorally once before training and four times after training through 14 to 16 days.

Outcome measures

We will assess homosynaptic depression of the soleus H reflex (an expression of the excitability of the alpha-motorneuron pool), a phenomenon that is not susceptible to descending suprasegmental influences but depends on the history of information arriving to the alpha-motorneuron from the periphery. Amount of homosynaptic depression will be correlated with the behavioral learning assessed by improvement in control of stepping speed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers (age 21 to 65 years) who are willing to participate and who are considered able to cylce for 16 minutes based on neurological and physical exams will be eligible for the study. Reproductive age women with a negative pregnancy test.

EXCLUSION CRITERIA:

Subjects with history of heart condition, unresponsive arterial hypertension, diabetes, chronic back pain, sciatica, peripheral neuropathy, rheumatoid arthritis, active joint deformity of arthritic origin, alcohol or drug abuse, psychiatric disorder requiring hospitalization or prolonged treatment, head injury with loss of consciousness, epilepsy. Subjects with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system or disorders of the blood coagulation system. Pregnant women.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-12-01; Study Completion 2008-05-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Faist M, Mazevet D, Dietz V, Pierrot-Deseilligny E. A quantitative assessment of presynaptic inhibition of Ia afferents in spastics. Differences in hemiplegics and paraplegics. Brain. 1994 Dec;117 ( Pt 6):1449-55. doi: 10.1093/brain/117.6.1449. PMID 7820579